CLINICAL TRIAL: NCT07096687
Title: Targeted Temperature Management for Neuroprotection in Acute Ischemic Stroke: A Randomized Controlled Pilot Trial
Brief Title: Targeted Temperature Management in Acute Ischemic Stroke
Acronym: TTM-STROKE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Usl di Bologna (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TTM-STROKE
Record Dates: First submitted 2025-07-24; First posted 2025-07-31 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Ischemic Stroke
Keywords: ischemic stroke; neuroprotection; targeted temperature management
MeSH Terms: conditions — Ischemic Stroke | interventions — Hypothermia, Induced

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): Patients will receive targeted temperature management to maintain normothermia using the CB240_Aurora device.
  Interventions: Device: Targeted Temperature Management with CB240_Aurora; Device: Standard of care Temperature treatment
- Control Arm (Sham Comparator): CB240_Aurora device used exclusively in temperature monitoring and control mode according to clinical standards
  Interventions: Device: Standard of care Temperature treatment

INTERVENTIONS:
Device: Targeted Temperature Management with CB240_Aurora — The proposed experimental treatment with the CB240_Aurora device will serve as a complementary approach to standard therapies, aiming to enhance their effectiveness. The device will continuously monitor body temperature and deliver treatment to maintain normothermia, defined as a temperature ≥36°C and <37°C at the time of study inclusion.
  Arms: Intervention Arm
Device: Standard of care Temperature treatment — In the control group, patients will receive treatment according to the latest guidelines for the management of ischemic stroke, including standard body temperature management. The CB240_Aurora device will be used exclusively in monitoring mode, without delivering any active treatment, and will be maintained for 72 consecutive hours from the time of enrollment

SUMMARY:
The goal of this interventional trial is to evaluate whether the CB240_Aurora medical device is effective for targeted temperature management in adult patients with acute ischemic stroke. The main questions it aims to answer are: Is the CB240_Aurora effective in maintaining normothermia in patients with acute ischemic stroke? Does the medical device improve clinical and radiological outcomes? Is the medical device well tolerated by patients? Researchers will compare an interventional arm, in which the CB240_Aurora measures and treats body temperature to maintain normothermia, with a control arm, in which the CB240_Aurora only measures but does not treat body temperature. Participants will wear the medical device for 72 consecutive hours in the Stroke Unit. Outcome assessments will be performed at 72 hours, 7 days, and 3 months.

DETAILED DESCRIPTION:
Neuroprotection is a potential therapeutic strategy to complement reperfusion and prevent the progression of cerebral ischemia in patients with acute ischemic stroke. One of the most promising approaches is Targeted Temperature Management (TTM), which involves controlling body temperature to prevent fever, maintain normothermia, or induce hypothermia in order to reduce brain injury and improve clinical outcomes. While hypothermia has demonstrated clinical benefits in patients with cardiac arrest and hypoxic- schemic encephalopathy, no significant evidence currently supports its efficacy in acute stroke. Maintaining normothermia through TTM may offer similar neuroprotective benefits with fewer complications. Current guidelines for patients with intracerebral hemorrhage, subarachnoid hemorrhage, and ischemic stroke recommend maintaining body temperature between 36°C and 37.5°C, ideally using automated control systems.

In this context, Neuron Guard has developed the CB240_Aurora device, which targets cerebral temperature through the vascular anatomy of the neck to enhance heat exchange. This system has shown potential in stabilizing brain temperature while maintaining systemic normothermia and reducing systemic side effects. Its use could be extended beyond intensive care settings to broader patient populations, both for managing fever episodes and for enhancing neuroprotection.

The experimental treatment with the CB240_Aurora device is designed as a complementary approach to standard therapies, aiming to improve their effectiveness. The device will continuously monitor body temperature and deliver treatment to maintain normothermia, defined as a temperature ≥36°C and <37°C at the time of study inclusion.

In the control group, patients will receive care according to the latest ischemic stroke treatment guidelines, including standard temperature management. In this group, the CB240_Aurora device will be used exclusively for temperature monitoring without providing active treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years;
* Both sexes;
* Diagnosis of acute ischemic stroke confirmed by clinical evaluation by a neurologist and neuroimaging (CT or brain MRI);
* Acute ischemic stroke with symptom onset within 48 hours;
* Anterior circulation stroke with evidence on neuroimaging (CT angiography) of occlusion of the middle cerebral artery in segments M1, M2, or M3;
* NIHSS score between 6 and 25;
* First clinical stroke;
* Axillary temperature ≥36°C and <37°C;
* Informed consent obtained for study participation.

Exclusion Criteria:

* Stroke involving multiple vascular territories;
* Presence of intracerebral hemorrhage;
* Pregnancy;
* Moderate-to-severe or severe pre-stroke disability defined as mRS >3;
* Presence of a cardiac pacemaker or any other conditions contraindicating brain MRI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2025-09-11 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Duration of normothermia maintenance during the first 72 hours | T0 (0 hour)T1; ( 72 hours)
  Measure the duration (in hours) of maintained normothermia (between >36°C and <37°C) through axillary temperature monitoring during the first 72 hours.

SECONDARY OUTCOMES:
Modified Rankin Scale (mRS) | T2 (day 7); T3 (day 90)
  Functional outcome at 3 months, defined as the Modified Rankin Scale (mRS) score ranging from 0 to 6, with higher scores indicating worse outcomes
National Institutes of Health Stroke Scale (NIHSS) | T2 (day 7); T3 (day 90)
  Clinical outcome at 7 days, defined as the National Institutes of Health Stroke Scale (NIHSS) score ranging from 0 to 42, with higher scores indicating worse outcomes
Change in the volume of the ischemic lesion measured by MRI | T2 (day 7)
  Ischemic lesion volume will be evaluated by MRI at day 7 from randomization (T0)
hemorrhagic transformation of the ischemic lesion at MRI | T2 (day 7)
  hemorrhagic transformation of the ischemic lesion at MRI
Incidence of adverse events (AEs) and severe AEs (SAEs) that are related to treatment. | T0 (day 0); T1 (day 3); T2 (day 7); T3( day 90)
  Safety will be assessed by measuring the incidence of AEs and SAEs throughout the stimulation period and during the 3-month follow-up
Number of patients requiring to stop treatment sessions | from T0 (day 0); T3 (day 90)
Qualitative assessment of device tollerability (QADT) | T2 (day 7); T3 (day 90)
  An ad hoc questionnaire to assess the tolerability of the device (e.g., nausea, headache, palpitations, anxiety, sweating) will be administered daily during the entire hospital stay and, after discharge, at each outpatient follow-up visit. Responses will be categorized as: Response No (Better Outcome) and Response Yes (Worse Outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Zini, Principal Investigator — IRCCS Istituto delle Scienze Neurologiche di Bologna - AUSL of Bologna
Locations (1):
- IRCCS Istituto delle Scienze Neurologiche di Bologna - AUSL of Bologna, Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lavinio A, Beqiri E, Kataria K. A Novel Technology for Targeted Brain Temperature Management. Neurocrit Care. 2024 Apr;40(2):785-790. doi: 10.1007/s12028-023-01800-7. Epub 2023 Jul 27. No abstract available. PMID 37498461
- [Background] Lavinio A, Andrzejowski J, Antonopoulou I, Coles J, Geoghegan P, Gibson K, Gudibande S, Lopez-Soto C, Mullhi R, Nair P, Pauliah VP, Quinn A, Rasulo F, Ratcliffe A, Reddy U, Rhodes J, Robba C, Wiles M, Williams A. Targeted temperature management in patients with intracerebral haemorrhage, subarachnoid haemorrhage, or acute ischaemic stroke: updated consensus guideline recommendations by the Neuroprotective Therapy Consensus Review (NTCR) group. Br J Anaesth. 2023 Aug;131(2):294-301. doi: 10.1016/j.bja.2023.04.030. Epub 2023 May 22. PMID 37225535
- [Background] Dankiewicz J, Cronberg T, Lilja G, Jakobsen JC, Levin H, Ullen S, Rylander C, Wise MP, Oddo M, Cariou A, Belohlavek J, Hovdenes J, Saxena M, Kirkegaard H, Young PJ, Pelosi P, Storm C, Taccone FS, Joannidis M, Callaway C, Eastwood GM, Morgan MPG, Nordberg P, Erlinge D, Nichol AD, Chew MS, Hollenberg J, Thomas M, Bewley J, Sweet K, Grejs AM, Christensen S, Haenggi M, Levis A, Lundin A, During J, Schmidbauer S, Keeble TR, Karamasis GV, Schrag C, Faessler E, Smid O, Otahal M, Maggiorini M, Wendel Garcia PD, Jaubert P, Cole JM, Solar M, Borgquist O, Leithner C, Abed-Maillard S, Navarra L, Annborn M, Unden J, Brunetti I, Awad A, McGuigan P, Bjorkholt Olsen R, Cassina T, Vignon P, Langeland H, Lange T, Friberg H, Nielsen N; TTM2 Trial Investigators. Hypothermia versus Normothermia after Out-of-Hospital Cardiac Arrest. N Engl J Med. 2021 Jun 17;384(24):2283-2294. doi: 10.1056/NEJMoa2100591. PMID 34133859
- [Background] Wang H, Olivero W, Lanzino G, Elkins W, Rose J, Honings D, Rodde M, Burnham J, Wang D. Rapid and selective cerebral hypothermia achieved using a cooling helmet. J Neurosurg. 2004 Feb;100(2):272-7. doi: 10.3171/jns.2004.100.2.0272. PMID 15086235
- [Background] Lyden P, Hemmen T, Grotta J, Rapp K, Ernstrom K, Rzesiewicz T, Parker S, Concha M, Hussain S, Agarwal S, Meyer B, Jurf J, Altafullah I, Raman R; Collaborators. Results of the ICTuS 2 Trial (Intravascular Cooling in the Treatment of Stroke 2). Stroke. 2016 Dec;47(12):2888-2895. doi: 10.1161/STROKEAHA.116.014200. Epub 2016 Nov 10. PMID 27834742
- [Background] Lyden PD, Allgren RL, Ng K, Akins P, Meyer B, Al-Sanani F, Lutsep H, Dobak J, Matsubara BS, Zivin J. Intravascular Cooling in the Treatment of Stroke (ICTuS): early clinical experience. J Stroke Cerebrovasc Dis. 2005 May-Jun;14(3):107-14. doi: 10.1016/j.jstrokecerebrovasdis.2005.01.001. PMID 17904009
- [Background] You JS, Kim JY, Yenari MA. Therapeutic hypothermia for stroke: Unique challenges at the bedside. Front Neurol. 2022 Oct 3;13:951586. doi: 10.3389/fneur.2022.951586. eCollection 2022. PMID 36262833
- [Background] Yenari MA, Han HS. Neuroprotective mechanisms of hypothermia in brain ischaemia. Nat Rev Neurosci. 2012 Feb 22;13(4):267-78. doi: 10.1038/nrn3174. PMID 22353781
- [Background] Edwards AD, Brocklehurst P, Gunn AJ, Halliday H, Juszczak E, Levene M, Strohm B, Thoresen M, Whitelaw A, Azzopardi D. Neurological outcomes at 18 months of age after moderate hypothermia for perinatal hypoxic ischaemic encephalopathy: synthesis and meta-analysis of trial data. BMJ. 2010 Feb 9;340:c363. doi: 10.1136/bmj.c363. PMID 20144981
- [Background] Hypothermia after Cardiac Arrest Study Group. Mild therapeutic hypothermia to improve the neurologic outcome after cardiac arrest. N Engl J Med. 2002 Feb 21;346(8):549-56. doi: 10.1056/NEJMoa012689. PMID 11856793
- [Background] Bernard SA, Gray TW, Buist MD, Jones BM, Silvester W, Gutteridge G, Smith K. Treatment of comatose survivors of out-of-hospital cardiac arrest with induced hypothermia. N Engl J Med. 2002 Feb 21;346(8):557-63. doi: 10.1056/NEJMoa003289. PMID 11856794
- [Background] Reith J, Jorgensen HS, Pedersen PM, Nakayama H, Raaschou HO, Jeppesen LL, Olsen TS. Body temperature in acute stroke: relation to stroke severity, infarct size, mortality, and outcome. Lancet. 1996 Feb 17;347(8999):422-5. doi: 10.1016/s0140-6736(96)90008-2. PMID 8618482
- [Background] Madden LK, Hill M, May TL, Human T, Guanci MM, Jacobi J, Moreda MV, Badjatia N. The Implementation of Targeted Temperature Management: An Evidence-Based Guideline from the Neurocritical Care Society. Neurocrit Care. 2017 Dec;27(3):468-487. doi: 10.1007/s12028-017-0469-5. PMID 29038971
- [Background] Donnan GA, Davis SM, Parsons MW, Ma H, Dewey HM, Howells DW. How to make better use of thrombolytic therapy in acute ischemic stroke. Nat Rev Neurol. 2011 Jun 14;7(7):400-9. doi: 10.1038/nrneurol.2011.89. PMID 21670766
- [Background] Savitz SI, Baron JC, Yenari MA, Sanossian N, Fisher M. Reconsidering Neuroprotection in the Reperfusion Era. Stroke. 2017 Dec;48(12):3413-3419. doi: 10.1161/STROKEAHA.117.017283. Epub 2017 Nov 16. No abstract available. PMID 29146878
- [Background] Rabinstein AA, Albers GW, Brinjikji W, Koch S. Factors that may contribute to poor outcome despite good reperfusion after acute endovascular stroke therapy. Int J Stroke. 2019 Jan;14(1):23-31. doi: 10.1177/1747493018799979. Epub 2018 Sep 6. PMID 30188259
- [Background] Vanacker P, Lambrou D, Eskandari A, Mosimann PJ, Maghraoui A, Michel P. Eligibility and Predictors for Acute Revascularization Procedures in a Stroke Center. Stroke. 2016 Jul;47(7):1844-9. doi: 10.1161/STROKEAHA.115.012577. Epub 2016 Jun 14. PMID 27301945
- [Background] Powers WJ. Acute Ischemic Stroke. N Engl J Med. 2020 Jul 16;383(3):252-260. doi: 10.1056/NEJMcp1917030. No abstract available. PMID 32668115
- [Background] Feigin VL, Forouzanfar MH, Krishnamurthi R, Mensah GA, Connor M, Bennett DA, Moran AE, Sacco RL, Anderson L, Truelsen T, O'Donnell M, Venketasubramanian N, Barker-Collo S, Lawes CM, Wang W, Shinohara Y, Witt E, Ezzati M, Naghavi M, Murray C; Global Burden of Diseases, Injuries, and Risk Factors Study 2010 (GBD 2010) and the GBD Stroke Experts Group. Global and regional burden of stroke during 1990-2010: findings from the Global Burden of Disease Study 2010. Lancet. 2014 Jan 18;383(9913):245-54. doi: 10.1016/s0140-6736(13)61953-4. PMID 24449944